CLINICAL TRIAL: NCT06004960
Title: An Open-Label, Phase 1 Study in Healthy Volunteers to Evaluate the Mass Balance Recovery and Metabolic Disposition of a Single Oral Dose of [14C]CCX168
Brief Title: A Study to Assess the Mass Balance Recovery (Absorption, Distribution, Metabolism and Excretion) of [14C]CCX168 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CL004_168
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Anti-neutrophil Cytoplasmic Antibody-associated Vasculitis
Keywords: Vasculitis; Complement; C5aR; Vascular diseases; Cardiovascular diseases; Systemic lupus erythematosus
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis; Vascular Diseases; Cardiovascular Diseases; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]CCX168 (Experimental): Participants will receive a single oral dose of [14C]CCX168 100 mg containing 400 μCi of [14C] on Day 1.
  Interventions: Drug: [14C]CCX168

INTERVENTIONS:
Drug: [14C]CCX168 — Administered orally.

SUMMARY:
The primary objective of this study is to perform mass balance following a single oral dose of [14C]CCX168 in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

* Males, aged 18-55 years inclusive, who are in generally good health, whose body mass index is 19.0 to 30.0 kg/m^2 inclusive;
* Willing and able to give written Informed Consent and to comply with the requirements of the study protocol;
* Negative result of the human immunodeficiency virus screen, the hepatitis B screen, and the hepatitis C screen;
* Judged to be healthy by the Investigator, based on medical history, physical examination (including electrocardiogram), and clinical laboratory assessments. Participants with clinical laboratory values that are outside of normal limits and/or with other abnormal clinical findings that are judged by the Investigator not to be of clinical significance may be entered into the study;
* Male participants with partners of childbearing potential may participate if adequate contraception is used during, and for 90 days after, any administration of study medication;
* Males must refrain from sperm donation for 90 days following completion of the study;
* Participants must have regular (at least once per day) bowel movements.

Exclusion Criteria:

* Participated in any studies where any radiolabeled drug was administered in the year prior to enrollment;
* Received a diagnostic or therapeutic radiation dose (such as a barium meal, serial x-ray scan, or computed tomography scan) within 1 year of enrollment or are currently employed in a job requiring radiation exposure monitoring;
* Expected requirement for use of any medication during the study period;
* For at least 3 days prior to enrollment and throughout the blood sample collection period, participants will not be allowed to eat any food or drink any beverage containing alcohol, caffeine, grapefruit, grapefruit juice, Seville oranges, or charbroiled meat;
* History within the three months prior to study entry of use of tobacco and/or nicotine containing products;
* History within one year prior to study entry of illicit drug use;
* History of alcohol abuse at any time in the past;
* History of any form of cancer;
* History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the participant at unacceptable risk for study participation;
* Donated or lost more than 350 mL of blood or blood products within 56 days prior to screening, or donated plasma within 7 days of dosing;
* Participant's hemoglobin less than 12 g/dL, confirmed by repeat measurement;
* Participated in any clinical study of an investigational product within 30 days prior to dosing;
* Participant has any evidence of hepatic disease; aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, or bilirubin greater than the upper limit of normal, unless considered not clinically significant by the Investigator;
* Participant's white blood cell count is below the lower limit of normal at Screening or Check-in (Day -1), confirmed by repeat measurement;
* Participant has any evidence of renal impairment; serum creatinine greater than the upper limit of normal, unless considered not clinically significant by the investigator;
* Participant's urine tested positive at Screening and/or on Study Day -1 for any of the following: opioids, amphetamines and methamphetamines, cannabinoids, benzodiazepines, barbiturates, cocaine, cotinine, ecstasy, methadone, phencyclidine, tricyclic antidepressants, or alcohol Breathalyzer test allowed for alcohol).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy adult males will be enrolled.
Enrollment: 6 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

PRIMARY OUTCOMES:
Cumulative Percentage of the Administered Dose of [14C]CCX168 Recovered in Urine | Up to Day 15
Cumulative Percentage of the Administered Dose of [14C]CCX168 Recovered in Feces | Up to Day 15

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Time of Occurrence of Maximum Observed Concentration (Tmax) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Elimination Rate Constant (λz) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Apparent Terminal Half-life (t½z) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Apparent Total Clearance (CL/F) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Apparent Volume of Distribution (Vz/F) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Area Under the Concentration-Time Curve from Time 0 to Time t (AUC0-t) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUCinf) of Total Radioactivity in Plasma and Whole Blood | Up to Day 10
Area Under the Concentration-Time Curve from Time 0 to 24 Hours (AUC0-24) of Total Radioactivity in Plasma and Whole Blood | Up to 24 hours
Cmax of CCX168 and Metabolites in Plasma | Up to Day 10
Tmax of CCX168 and Metabolites in Plasma | Up to Day 10
λz of CCX168 and Metabolites in Plasma | Up to Day 10
t½z of CCX168 and Metabolites in Plasma | Up to Day 10
CL/F of CCX168 and Metabolites in Plasma | Up to Day 10
Vz/F of CCX168 and Metabolites in Plasma | Up to Day 10
AUC0-t of CCX168 and Metabolites in Plasma | Up to Day 10
AUCinf of CCX168 and Metabolites in Plasma | Up to Day 10
AUC0-24 of CCX168 and Metabolites in Plasma | Up to 24 hours
Percentage of Unchanged [14C]CCX168 Recovered in Urine, Feces, and Vomitus | Up to Day 15
Percentage of [14C]-Metabolite Recovered in Urine, Feces, and Vomitus | Up to Day 15
Amount of Unchanged [14C]CCX168 Recovered in Urine, Feces, and Vomitus (Auinf + Afinf + Avinf) | Up to Day 15
Amount of [14C]-Metabolite Recovered in Urine, Feces, and Vomitus (Amxuinf + Amxfinf + Amxvinf) | Up to Day 15
Renal Clearance (CLR) of [14C]CCX168 | Up to Day 15
Renal Clearance of [14C]-Metabolite (CLRmx) | Up to Day 15
Number of Participants Experiencing Adverse Events (AEs) | Up to Day 29
Number of Participants Experiencing Clinically Significant Changes in Laboratory Parameters | Up to Day 29
Number of Participants Experiencing Clinically Significant Changes in Vital Sign Parameters | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com